CLINICAL TRIAL: NCT02839317
Title: Comparison of Fecal Microbiota Between Patients With Early and Late Crohn's Disease and Relationship With Different Genetic and Serological Profiles
Brief Title: COmparison of MicroBiota AccordIng to Age in Crohn's Disease (COMeBACk)
Acronym: COMeBACk
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_71; 2014-A01225-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease
Keywords: Dysbiosis; Crohn's disease; Age
MeSH Terms: conditions — Crohn Disease; Dysbiosis | interventions — Biological Products

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples Blood samples (DNA extraction) and sera Salivary samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Biological in pediatric CD: 75 pediatric-onset CD Biological
  Interventions: Biological: Biological
- Biological in pediatric controls: 75 pediatric controls matched on gender, age and area of residence Biological
  Interventions: Biological: Biological
- Biological in elderly CD: 75 elderly-onset CD Biological
  Interventions: Biological: Biological
- Biological in elderly controls: 75 elderly controls matched on gender, age and area of residence Biological
  Interventions: Biological: Biological

INTERVENTIONS:
Biological: Biological — comparison of microbiota, genetic profile between pediatric- and elderly-onset CD
  Other Names: Dysbiosis

SUMMARY:
The cause of CD could be different according to age at onset of CD symptoms. Indeed we know that some very young patients at CD diagnosis have particular genetic variants as abnormalities of the IL10R that are regarded as quite monogenic disease. In the other way, the microbiota also undergoes substantial changes at the extremes of life, in infants and older people and the ramifications of which are very few being explored. The comparison of microbiota by principal component analysis and genetic profile of patients with CD beginning at the extremes of life could help us to better known physiopathology of CD according to age and provide arguments that CD beginning at the extremes of life could be different diseases.

The aim of the study is to ascertain through population-based study the hypothesis that gut microbiota is different between paediatric-onset and elderly-onset CD patients in relation with genetic and environmental mechanisms. The results will provide a better knowledge of the etiopathogenic ways in CD and propose a personalized therapeutic care based on age at CD onset (i.e. according to the gut bacteria involved).

DETAILED DESCRIPTION:
The primary aim is to describe by principal component analysis and compare the gut microbiota between subgroups of paediatric-onset (n=75), elderly-onset CD patients (n=75) and control subjects (75 paediatric control and 75 elderly control subjects matched on age) without an a priori approach of high throughput sequencing of bacterial DNA. As it has been shown that the type of IBD-associated dysbiosis depends on ileal involvement, Paediatric-onset and elderly-onset CD patients will be stratified according this parameter.

The secondary aims are:

* (I) Find specific bacteria involved in paediatric- and elderly-onset patients using PLS Discriminant Analysis (PLS-DA) that is a classical PLS regression (with a regression mode) but where the response variable is categorical.
* (II) Search for an association between bacterial dysbiosis and different genetic backgrounds in patients according to age at CD onset (paediatric-onset vs elderly-onset) and in control subjects;
* (III) Quantify of bacteria with invasive properties (E. coli, including adherent-invasive E.coli, Shigella, Salmonella, Yersinia, Campylobacter), and fecal fungal flora (Candida albicans, in particular) and their association with genetic and serological profiles according to age at CD onset and in control subjects; this study will include the comparison of the gut microbiome between subgroups of paediatric-onset, elderly-onset CD patients and control subjects.
* (IV) Study of environmental risk factors using a questionnaire to be submitted to CD patients and control subjects.

The results would provide a better knowledge of the etiopathogenic ways in CD and would downstream open the way towards clinical trials focused on specific microbiota disorders according to age at CD onset. This project will help to decipher the potential involvement of specific bacteria in the physiopathology of CD. This could lead to the development of new therapeutic strategies either using optimized current treatments targeting bacteria. Data from clinical trials which for the great majority rarely include paediatric patients and set an upper limit for study eligibility at 65 years of age are thus focusing on adult-onset disease. Thus the potential specificities of paediatric- and elderly-onset diseases are not taken into account. A better knowledge of characteristics of CD at the extreme of life will be important to set up innovative clinical trials including specific therapeutics adapted to patients where disease occurred at the extreme age of life, especially as these patients did not benefited of specific trials. The ultimate goal is a better quality of care delivered to paediatric- and elderly-onset CD patients.

ELIGIBILITY:
Inclusion Criteria:

* CD patients Patients aged less than 17 years (paediatric-CD group) or more than 40 years (elderly-CD group) at definite or probable CD diagnosis, defined according to Epimad's criteria2,4.

CD diagnosis within 5 years prior inclusion. Patients with CD in remission with or without corticosteroids, 5-ASA or nutrition.

Agreeing to participate in the project and have signed consent, Being insured

* Control subjects Patients aged less than 17 years (paediatric-control group) or more than 40 years (elderly-control group) Agreeing to participate in the project and have signed consent, Being insured

Exclusion Criteria:

* Pregnant or lactating Subject who underwent bowel resection Subject taking antibiotics, prebiotics, probiotics or bowel preparation in 6 weeks sampling seat will be temporarily suspended. The sampling will be done remotely and delayed (> 6 weeks) of treatment discontinuation or antibiotic bowel preparation.

A person taking or have taken a topical treatment within 6 weeks before inclusion Persons who have undergone surgical resection Nobody emergency Topic guardianship, curator ship or judicial protection, persons deprived of liberty Subject does not speak French Subject unable to answer questions or express

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric- onset (n=75), elderly-onset CD patients (n=75) and control subjects matched on age, gender and geographical origin (urban, periurban and rural area according to INSEE data) in each group (n=150) will be recruited through a large population-based registry of IBD patients (EPIMAD Registry). In 2 case-control studies, controls (n=150) will be matched to cases by age (± 2 years), gender and geographical origin (urban, periurban and rural area according to INSEE data). Control subjects will be recruited through paediatric and geriatric consultations in Lille University Hospital.
  The duration of recruitment will be 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Analysis of microbiota | 1 YEAR
  To describe by principal component analysis and compare the gut microbiota between subgroups of paediatric-onset (n=75), elderly-onset CD patients (n=75) and controls (150).

SECONDARY OUTCOMES:
Specific bacteria | 1 YEAR
  Find specific bacteria involved in paediatric- and elderly-onset patients using PLS Discriminant Analysis (PLS-DA)
Association between bacterial dysbiosis and different genetic backgrounds | 1 YEAR
  Search for an association between bacterial dysbiosis and different genetic backgrounds in patients according to age at CD onset (paediatric-onset vs elderly-onset) and in controls
Presence of bacteria with invasive properties (E. coli, including adherent-invasive E.coli, Shigella, Salmonella, Yersinia, Campylobacter), and fecal fungal flora (Candida albicans, in particular) | 1 YEAR
  Quantify of bacteria with invasive properties (E. coli, including adherent-invasive E.coli, Shigella, Salmonella, Yersinia, Campylobacter), and fecal fungal flora (Candida albicans, in particular)
Environmental risk factors | 1 YEAR
  Study of environmental risk factors using a questionnaire to be submitted to CD patients and controls .

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Gower-Rousseau, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (5):
- France (5):
  - Amiens University & Hospital, Amiens
  - Lille Hôpital Huriez, Lille
  - Lille Jean de Flandre Hospital, Lille
  - Lille University Hospital & EPIMAD Registry, Lille
  - Rouen University & Hospital, Rouen

IPD SHARING:
Plan to Share IPD: Undecided